CLINICAL TRIAL: NCT06232057
Title: The Effect of Preoperative Virtual Reality Glasses Use on Postoperative Pain and Anxiety in Women Having a Caesarean Section
Brief Title: Use of Virtual Reality Glasses for Pain and Anxiety After Cesarean
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Amasya University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: AmasyaÜ-Ketenedis-001
Record Dates: First submitted 2024-01-22; First posted 2024-01-30 (Actual); Last update posted 2024-10-18 (Actual); Status verified 2024-10

CONDITIONS: Cesarean Section; Pain, Postoperative; Anxiety
Keywords: Cesarean Section; Pain; Anxiety; Virtual reality
MeSH Terms: conditions — Pain, Postoperative; Anxiety Disorders; Pain

STUDY DESIGN:
Intervention Model Description: This randomized controlled study will be conducted with women who had a cesarean in the Obstetrics and Gynecology clinic of a public hospital in northern Turkey.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): Virtual Reality Application Group
  Interventions: Other: Virtual Reality
- Control Group (No Intervention): Control group without any intervention

INTERVENTIONS:
Other: Virtual Reality — Women in the intervention group will be given a pre-test (STAI) before cesarean. Then, they will be shown a relaxing video (video with nature views accompanied by nature sounds) through virtual reality glasses for a maximum of 20 minutes. After a cesarean, women's anxiety levels (STAI) will be evaluated within the first 4 hours postoperatively. Pain levels (VAS) will be assessed postoperatively at the 2nd, 4th, and 6th hours.
  Arms: Intervention Group

SUMMARY:
The goal of this randomized controlled trial is to examine the effect of preoperative virtual reality used before cesarean on postoperative pain and anxiety. The main question[s] it aims to answer are:

* What is the anxiety level of women in the intervention and control groups after using virtual reality?
* What is the pain level of women in the intervention and control groups after using virtual reality?

Women in the intervention group will be shown a relaxing video accompanied by virtual reality glasses before cesarean. No intervention will be applied to women in the control group. Researchers will compare pre- and post-operative anxiety levels and post-operative pain levels of both groups.

DETAILED DESCRIPTION:
Cesarean is a major surgical operation that is widely performed around the world. Pain after cesarean is more significant than expected, and pain control remains a problem. In addition, the women undergoing cesarean experience stress and anxiety due to the surgical process. Anxiety and pain experienced after cesarean affect the mother physiologically and psychologically, negatively affecting the healing process. Therefore, it is essential to determine interventions that will reduce pain and anxiety in women undergoing cesarean. This study aims to examine the effect of preoperative virtual reality use on postoperative pain and anxiety in women undergoing cesarean.

This study has a randomized controlled experimental design. The research will be carried out in the Obstetrics and Gynecology Clinic of a public hospital in the North of Turkey. Women who had a cesarean will be included in the study. Participants will be randomly assigned to the intervention or control group using a computer-generated list. A data collection form including an Introductory information form including sociodemographic and obstetric characteristics, Spielberger State-Trait Anxiety Inventory (STAI), and Visual Analog Scale (VAS) will used for each participant. After obtaining written informed consent, the anxiety levels of women in the intervention and control groups will be determined by applying a pre-test (STAI). Then, the women in the intervention group will be shown a relaxing video (video with a nature view accompanied by nature sounds) through preoperative virtual reality glasses. No intervention will be applied to women in the control group. After surgery, the anxiety levels of women in both groups will be evaluated in the first 4 hours, and the pain levels will be evaluated in the 2nd, 4th, and 6th hours. The IBM SPSS (Statistical Package for the Social Sciences) 21.0 package program will be used to evaluate the data obtained in the study.

ELIGIBILITY:
Inclusion Criteria:

* 18 years and over
* Communicate in Turkish
* Must have cesarean with spinal anesthesia
* Must have cesarean after the 37th week of pregnancy
* Must have a planned cesarean

Exclusion Criteria:

* Under 18 years
* Not being able to speak Turkish
* Vision and hearing problem
* Cesarean section with general anesthesia
* Emergency cesarean

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2024-02-01 (Actual); Primary Completion 2024-07-10 (Actual); Study Completion 2024-07-10 (Actual)

PRIMARY OUTCOMES:
Preoperative anxiety level | Preoperatif
  Preoperative anxiety level will be measured with STAI.
Postoperative pain level-1 | Postoperative 2nd hour
  The pain level at the 2nd hour after cesarean section will be measured with VAS.
Postoperative anxiety level | Within the first 4 hours postoperatively
  Anxiety level after cesarean section will be measured with STAI within the first 4 hours.
Postoperative pain level-2 | Postoperative 4th hour
  The pain level at the 4th hour after cesarean section will be measured with VAS.
Postoperative pain level-3 | Postoperative 6th hour
  The pain level at the 6th hour after cesarean section will be measured with VAS.

CONTACTS AND LOCATIONS:
Overall Officials: ELİF KETEN EDİS, Study Director — Amasya University
Locations (1):
- Amasya University, Amasya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No